CLINICAL TRIAL: NCT06123013
Title: Music Therapy in Patients Undergoing Pancreatic Surgery (MUSIC PUPS): A Mixed Methods Feasibility Study
Brief Title: Music Therapy in Patients Undergoing Pancreatic Surgery (MUSIC PUPS)
Acronym: MUSIC PUPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Samuel Rodgers-Melnick, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY20221489
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Whipple Procedure; Distal Pancreatectomy; Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music assisted relaxation (Experimental): Participants will receive a tailored music-assisted relaxation and imagery intervention
  Interventions: Behavioral: Music Assisted Relation Intervention (MARI)

INTERVENTIONS:
Behavioral: Music Assisted Relation Intervention (MARI) — A standardized 30-minute MARI intervention, personalized to the participant's music and imagery preferences. During the MARI intervention, the board certified music therapist (MT-BC) will provide live guitar accompaniment personalized to the participant's music preferences and read from a standardized script directing the participant to relax muscles of the body, practice deep breaths, and explore a relaxing place.

SUMMARY:
Pilot single arm non-randomized trial to determine the feasibility and acceptability of: 1) a tailored music-assisted relaxation and imagery intervention; 2) biological sample collection; and 3) mobile device patient-reported outcome (MDPRO) collection in adults hospitalized for pancreatic surgery experiencing acute pain.

DETAILED DESCRIPTION:
After the participant's pancreatic surgery and during their post-surgery hospitalization, the RA will confirm participant eligibility and continued willingness to participate. About an hour later, the RA will return to the participant's room. Before collecting any data, the RA will ask the participant if their pain will permit them to continue and if they would like to proceed. If the participant responds affirmatively, the RA will document this in REDCap and then will proceed to collect baseline (Time 0) patient-reported outcomes (PROs) (i.e., 0-10 ratings of pain, stress, and anxiety) using a REDCap instrument administered on an iPad. The RA will not view the participant's PRO responses. If the participant is currently utilizing a patient-controlled analgesia (PCA) pump, the RA will collect measures of medication usage from the PCA pump. The RA will also collect a peripheral blood sample using a Spot On Sciences HemaSpot-HF. The research team chose the HemaSpot HF because it is an efficient and less invasive means of collecting capillary blood. Using the HemaSpot HF also poses less risk and discomfort to these patients who recently underwent major surgery. Following baseline measure collection, the RA will leave the participant's room.

Following Time 0, the MT-BC will deliver a standardized 30-minute MARI intervention, personalized to the participant's music and imagery preferences. Prior to the intervention, the MT-BC will verify the participant's music and imagery preferences discussed with the RA earlier in the day. During the MARI intervention, the MT-BC will provide live guitar accompaniment personalized to the participant's music preferences and read from a standardized script directing the participant to relax muscles of the body, practice deep breaths, and explore a relaxing place. This intervention will be recorded live and exported to either a study iOS device (e.g., iPod touch, iPhone) programmed to track MARI recording use or uploaded to a Box folder that will be shared with the participant to listen to on their own device. Following the MARI intervention, the MT-BC will briefly process the participant's experience by asking them how the experience was for them and to describe in their own words how they are feeling after the MARI intervention. (please see the attachment "MUSIC PUPS Post MARI Debriefing" for more details). The RA will export the MARI recording to a Box folder that the participant can access using the iOS device.

Immediately following the MARI intervention and post-intervention processing, the MT-BC will leave the participant's room. The RA will then enter the participant's room again. The RA will confirm that the participant is not in too much pain to continue and would like to continue with study procedures, documenting this in REDCap, before collecting post-intervention PROs and peripheral blood smear measures (Time 1). After collecting these measures, the RA will wait in the participant's room for 15 minutes. At 15-minutes post-intervention (Time 2), the RA will again collect PROs and a final peripheral blood smear measure.

Then, the RA will show the participant how to access the MARI recording and enter MDPRO measurements using either the study iOS device or their own device. The RA will instruct the participant to listen to the MARI intervention 3x/day and complete 3 MDPRO measurements each day until discharge. The iOS device will be locked to the participant's tray table to prevent it from being lost or stolen during the participant's hospitalization.

Following the collection of blood samples and PROs, the RA will conduct a review of the participant's medical record to collect data on the participant's demographics, clinical characteristics, and pain medications administered pre-intervention. The RA will enter this data into REDCap. Following sample collection, blood samples will be temporarily stored within the Connor Whole Health research office. Samples will then be shipped within 12 hours to Manoj Bhasin's lab at Emory University for storage and subsequent analysis.

The RA will meet with each participant every day, Monday through Friday, until discharge to troubleshoot any barriers to MARI use or MDPRO collection. Each day, before any troubleshooting or collecting any data, the RA , like on day one, will (1) check in with the treating physician and/or the clinical nurse; (2) ask the participant if their pain level will permit them to participate; and (3) ask the participant if they still want to participate in study procedures. If the participant responds affirmatively to continuing study procedures, the RA will document this in REDCap and then proceed with troubleshooting and data collection. The RA will record any barriers to MARI use and/or MDPRO collection (i.e., forgot, technical difficulties, off the floor for a procedure) as well as the participant's self-reported use of MARI in the last 24 hours. From Day 2 (i.e., the day after the live MARI intervention) until the participant is discharged from the hospital, the participant will receive three notifications per day (i.e., morning, afternoon, and evening) on the iOS device to complete MDPRO measures. The participant's use of the MARI recording will be tracked using file utilization measures available within Box.com. No PHI will be entered into the Box.com folder. The RA will also track the participant's use of pain medications (recorded in the EHR or on the PCA). All data will be stored in REDCap.

On the day of the participant's discharge from the hospital, the RA will collect the study iOS device, if applicable. The RA will provide the participant with the MARI recording via email and a Box.com link to allow the participant to access the recording post-discharge. If desired, the RA will also provide the recording via a compact disk. Following discharge, the study coordinator will arrange a time for the participant to complete a semi-structured interview over Zoom. One to two weeks after the participant's discharge from the hospital, researchers will meet with the participant over a HIPAA-compliant commercial tele-health platform to complete a semi-structured interview. If the participant is expected to be discharged over the weekend, the RA will provide the MARI recording resources on the Friday before the weekend in which the participant is to be discharged.

Interview procedures Interviews will take place over a HIPAA-compliant commercial tele-health platform (i.e., Zoom for Healthcare) or over the phone one-to-two weeks after the participant is discharged from the hospital. During that interview, a researcher will ask the participant about their experience in the study and what they thought about the MARI intervention. The researcher conducting the interviews remotely will be in a private room when interviewing the participants and will be certified in human subject protection and GCP, researched credentialed if applicable, and on the study personnel table. The interview will take about 20 minutes and will be recorded and then transcribed by hand.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to speak and understand English
* Patient is scheduled to undergo a Whipple procedure or Distal pancreatectomy at UH Cleveland Medical Center with a standardized pain regimen
* Patient reports pain intensity of 4/10 or above on day 1 post-surgery

Exclusion Criteria:

* Subject has a significant visual impairment that has not been corrected
* Subject has a significant hearing impairment that has not been corrected
* Subject has a significant cognitive impairment that would prevent subject from participating in the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Delivery of a tailored music-assisted relaxation and imagery intervention (MARI) | Day 1 of the patients post pancreatic surgery hospital stay
  Percent of participants that complete the MARI intervention
Patient reported outcome (PRO) data collection | During the length of patient's hospital stay, up to two weeks
  Percent of completed patient reported outcomes surveys
Biological sample collection | Day 1 of patient's post pancreatic surgery hospital stay
  Percent of of viable biological samples collected

SECONDARY OUTCOMES:
Enrollment Rate | during the enrollment period of the study, up to two months
  enrolled participants as a percentage of those approached
Attrition Rate | While the study is active, up to 8 months
  percent of patients lost to follow up
Rate of MARI recording use | during patient's post pancreatic surgery hospital stay, up to two weeks
  MARI recording use as a percentage of expected usage

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Rodgers-Melnick, MPH, MT-BC, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT06123013/Prot_SAP_002.pdf
  • Informed Consent Form (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT06123013/ICF_003.pdf